CLINICAL TRIAL: NCT01280981
Title: A Multi-center, Open Label Extension Study to Evaluate the Safety of an Oral Dose of Tranexamic Acid (XP12B) Administered Three Times Daily During Menstruation for the Treatment of Menorrhagia
Brief Title: A Study of Tranexamic Acid (XP12B) in Women With Heavy Menstrual Bleeding
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Collaborators: Xanodyne Pharmaceuticals (Industry)
Responsible Party: Clinical Development Support, Ferring Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XP12B-MR-304
Record Dates: First submitted 2011-01-19; First posted 2011-01-21 (Estimated); Results first posted 2011-07-26 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2011-06

CONDITIONS: Menorrhagia
Keywords: Menorrhagia; Heavy Menstrual Bleeding; Lysteda
MeSH Terms: conditions — Menorrhagia | interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tranexamic acid (Experimental): Two 650 mg tablets orally 3 times per day with liquids for up to 5 days (not to exceed 3 doses in 1 day or 15 doses during the menstrual period).
  Interventions: Drug: Tranexamic acid

INTERVENTIONS:
Drug: Tranexamic acid — Tranexamic acid at an oral dose of 1.3 g administered 3 times per day for up to 5 days (maximum of 15 doses) during menstruation for 9 menstrual periods.
  Other Names: XP12B; Lysteda

SUMMARY:
This was a multicenter, open-label extension study for subjects completing either of 2 pivotal efficacy studies (NCT00401193 or NCT00386308). The study consisted of a treatment phase of 9 menstrual periods to assess the safety of tranexamic acid at an oral dose of 1.3 g administered 3 times per day for up to 5 days (maximum of 15 doses) during menstruation. After the last treatment period, a follow-up phone call occurred approximately 30 days (range 25 to 35 days) after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* The study enrolled subjects who had completed the double-blind therapy in either the XP12B-MR-301 or XP12B-MR-303 study, including scheduled evaluations, with no major protocol violations and no study events that, in the opinion of the investigator, would preclude the subject's entry into the open-label safety study.
* A negative urine pregnancy test was required immediately before entry into this study.
* Women must have been surgically sterile or, if of childbearing potential, must have been in a monogamous relationship with a sterile partner or a partner of the same sex.
* Women must have used an acceptable barrier contraception method with spermicide for the duration of the study or must have been using a copper intrauterine device (IUD).
* In the opinion of the investigator, the subject must be able to understand this study, cooperate with all study procedures, be able to return to the study site for visits within the required visit windows and be deemed likely to complete the study.
* Subject will provide voluntary, written consent to participate in the study by signing and dating an institutional review board (IRB)-approved informed consent before any procedures are performed or study drug is dispensed.

Exclusion Criteria:

* History or presence of clinically significant hepatic or renal disease or other medical disease that might confound the study or be detrimental to the subject (e.g., clinically significant cardiac arrhythmia, uncontrolled diabetes or uncontrolled hypertension) as determined by the investigator.
* Normal gynecological examination and breast examination.
* Clinically significant abnormalities on screening physical examination that might confound the study or be detrimental to the subject as assessed by the investigator. Abnormal clinically significant electrocardiograms (ECG) as determined by the centralized cardiologist, or laboratory tests suggestive of a potential pituitary-prolactin stimulating tumor (prolactin >=30 µg/L), thrombocytopenia (platelet count <100,000/mm3), uncontrolled hypothyroidism (TSH >=10 mU/L) or severe anemia (hemoglobin <8 g/dL]).
* Anovulatory dysfunctional uterine bleeding, metrorrhagia (irregular or frequent noncyclic flow), menometrorrhagia (irregular or frequent excessive noncyclic flow) or polymenorrhea (frequent flow, cycles of less than 21 days).
* History or presence of endometrial polyps, endometrial hyperplasia, endometrial carcinoma or cervical carcinoma (includes cervical carcinoma in situ).
* History of bilateral oophorectomy or hysterectomy.
* Women who are pregnant, breastfeeding, planning to become pregnant during the study or become pregnant during the study.
* History or active presence of myocardial infarction or ischemic disease. History or active presence of cerebrovascular accident, stroke, or transient ischemic attack.
* History or presence of thrombosis, thromboembolic disease or coagulopathy including, but not limited to, pulmonary embolism, deep venous thrombosis, phlebitis and any intravascular clotting disorder.
* History or known presence of acquired or inherited thrombophilia, including, but not limited to, antithrombin deficiency, Protein C and/or S deficiency, antiphospholipid deficiency, Factor V Leiden mutation and prothrombin mutation. Thalassemia or sickle cell disease (sickle cell trait individuals are not excluded).
* History or presence of subarachnoid hemorrhage.
* Use or anticipated use of medications taken to relieve β-Hydroxy β-methylbutyric acid (HMB) including the use of vaginal [rings, creams, gels] and transdermal hormone products; use of oral estrogen-, progestin- or SERM-containing drug products, or intrauterine progestins containing drug products. Use or anticipated use of Lupron (1 or 3 month) depot injection or estrogen pellet or long-acting progestin injectables.
* Use or anticipated use of meclofenamate sodium, mefenamic acid, danazol, or desmopressin acetate or herbal remedies. Herbal remedies include, but are not limited to, Capsella bursa pastoris (i.e. Sheperd's Purse), Agnus castus (i.e. Chasteberry, Vitex), Cimicifuga racemosa (i.e. Black Cohosh), Symphytum officionale (i.e. Comfrey), and/or Angelica sinensis (i.e. Dong Quai).
* Use of or anticipated use of the following drugs: oral, transdermal, injectable and vaginal ring (NuvaRing®) hormonal contraceptives; anticoagulants (warfarin [Coumadin®], heparin, low-molecular-weight heparin (LMWH), etc.), aminocaproic acid (Amicar®) or Plaquenil®.
* Current use of an intrauterine device (IUD) other than copper IUDs.
* History or presence of hypersensitivity or idiosyncratic reaction to antifibrinolytics (tranexamic acid or aminocaproic acid).
* Use of any investigational drug except XP12B-MR during the current study.
* Presence of untreated malabsorption disorder or malnutrition including, but not limited to, chronic diarrhea, celiac disease, short bowl syndrome, Whipple's disease or history of gastric bypass procedure.
* Presence of defective color vision as determined by the optometrist or ophthalmologist. Inability of the subject to correctly identify symbols on plate 7 of the HRR eye test is not considered defective color vision provided the subject correctly identifies the symbols on plates 11-20.
* History or presence of glaucoma, ocular hypertension, macular degeneration or retinopathies.
* History or presence of alcoholism or drug abuse within the past year.
* Malignancy, or treatment for malignancy, within the previous 2 years, with the exception of basal cell carcinomas of the skin or squamous cell carcinoma of the skin.
* Does not read or understand English.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 288 (Actual)
Dates: Start 2007-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (92):
- United States (92):
  - Radiant Research, Birmingham, Alabama
  - Women's Health Research, Phoenix, Arizona
  - Genova Clinical Research, Tucson, Arizona
  - Quality of Life Medical and Research Center, Tucson, Arizona
  - Radiant Research, Tucson, Arizona
  - Visions Clinical Research, Tucson, Arizona
  - Lynn Institute of the Ozarks, Little Rock, Arkansas
  - Searcy Medical Center, Searcy, Arkansas
  - Northern California Research Corp, Carmichael, California
  - Physicians' Research Options, LC, Lakewood, California
  - Sklar Center for Women's Wellness, Los Alamitos, California
  - Medical Center for Clinical Research, San Diego, California
  - INC Clinical Trials, Upland, California
  - Advanced Women's Health Institute, Denver, Colorado
  - Downtown Women's Health Care, Denver, Colorado
  - Nature Coast Clinical Research, Crystal River, Florida
  - University of Florida, Gainesville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - New Age Medical Research Corp, Miami, Florida
  - University of Miami Cedars Medical Center, Miami, Florida
  - Advanced Research Institute, New Port Richey, Florida
  - Segal Institute for Clinical Research, North Miami, Florida
  - Medical Network for Education & Research, Inc., Decatur, Georgia
  - The Women's Clinic, Boise, Idaho
  - Rosemark Womencare Specialists, Idaho Falls, Idaho
  - Provident Clinical Research, Bloomington, Indiana
  - Wichita Clinic, P.A., Newton, Kansas
  - Radiant Research, Overland Park, Kansas
  - York Clinical Consulting, Marrero, Louisiana
  - The Gynecology Center, Baltimore, Maryland
  - ClinSite, LLC, Ann Arbor, Michigan
  - Quest Research Institute, Bingham Farms, Michigan
  - Grand Valley Gynecologists PC, Grand Rapids, Michigan
  - Women's Health Care Specialist, Paw Paw, Michigan
  - KMED Research, Saint Clair Shores, Michigan
  - Center for Pharmaceutical Research, Kansas City, Missouri
  - Montana Medical Research, Inc, Missoula, Montana
  - The Women's Center of Western Nebraska, Scottsbluff, Nebraska
  - Office of R Garn Mabey, MD, Las Vegas, Nevada
  - Women's Health Research Center, LLC, Lawrenceville, New Jersey
  - Phoenix OB-GYN Assoc, LLC, Moorestown, New Jersey
  - American Clinical Trials, New York, New York
  - Duke Fertility Center, Durham, North Carolina
  - Women's Wellness Center, Durham, North Carolina
  - Lyndhurst Gynecologic Associates, Winston-Salem, North Carolina
  - Piedmont Medical Research Associates, Winston-Salem, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Triphase Research Ltd, Centerville, Ohio
  - Rapid Medical Research, Inc, Cleveland, Ohio
  - University Suburban Health Center, Cleveland, Ohio
  - Holzer Clinic, Gallipolis, Ohio
  - Physicians Research, Inc., Zanesville, Ohio
  - LION Research, Norman, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Clinical Trials of America, Eugene, Oregon
  - PMG/OB-GYN Health Center, Medford, Oregon
  - The Portland Clinic, Portland, Oregon
  - Abington Reproductive Medicine, PC, Abington, Pennsylvania
  - The Clinical Trial Center, Jenkintown, Pennsylvania
  - Family Medical Associates Research Dept, Levittown, Pennsylvania
  - Philadelphia Clinical Research, LLC, Philadelphia, Pennsylvania
  - University of Pennsylvania, Dept. OB/GYN, Philadelphia, Pennsylvania
  - Valley Forge OB/GYN, Phoenixville, Pennsylvania
  - Research Across America, Reading, Pennsylvania
  - Main Line OB/GYN, Strafford, Pennsylvania
  - Wexford Professional Bldg II, Wexford, Pennsylvania
  - SC Clinical Research Center, Columbia, South Carolina
  - Greenville Hospital System-Univ Med Group Dept, Greenville, South Carolina
  - Greenville Pharmaceutical Research, Greenville, South Carolina
  - Radiant Research, Greer, South Carolina
  - Seasons, Bristol, Tennessee
  - Southeastern Clinical Research, Chattanooga, Tennessee
  - Alpha Clinical Research, LLC, Clarksville, Tennessee
  - Volunteer Research Group, Knoxville, Tennessee
  - Research Memphis Associates, Memphis, Tennessee
  - Tennessee Women's Care, PC, Nashville, Tennessee
  - J&S Studies, Inc, College Station, Texas
  - OB/GYN Infertility & Preventive Medicine, Dallas, Texas
  - Phyllis Gee, MD, Plano, Texas
  - King's Daughters Clinic, Temple, Texas
  - Women's Healthcare, The Woodlands, Texas
  - Center of Reproductive Medicine, Webster, Texas
  - Mt. Timpanogos Women's Health Center, Pleasant Grove, Utah
  - Jean Brown Research, Salt Lake City, Utah
  - Physician's Research Options, Sandy City, Utah
  - Granger Medical OB/GYN, West Valley City, Utah
  - FAHC, Womens Health Research, Burlington, Vermont
  - Clinical Trials of Virginia, INC, Richmond, Virginia
  - Tidewater Clinical Research, Inc., Virginia Beach, Virginia
  - Valley Women's Clinic, Renton, Washington
  - North Spokane Women's Center, Spokane, Washington
  - Medical Associates Health Centers, Menomonee Falls, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who completed double-blind therapy in either study XP12B-MR-301 (NCT00401193) or XP12B-MR-303 (NCT00386308) could participate in this trial.
Period: Overall Study
Arm/Group | Tranexamic Acid
Started | 288
Intent to Treat (ITT) Population | 260 (Participants who took drug during at least one menstrual cycle)
Completed | 196
Not Completed | 92
Not completed — Withdrawal by Subject | 11
Not completed — Protocol Violation | 2
Not completed — Lack of Efficacy | 13
Not completed — Lost to Follow-up | 3
Not completed — Adverse Event | 6
Not completed — Irregular or discontinued menses | 3
Not completed — Failed to return | 45
Not completed — Non-compliance with protocol | 3
Not completed — Withdrawal of consent | 3
Not completed — Elective surgery | 2
Not completed — Study site closure | 1

BASELINE CHARACTERISTICS:
Arm/Group | Tranexamic Acid
Number analyzed (Participants) | 288
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 288
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 288
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Participants With Treatment-Emergent Adverse Events (AEs)
Description: Count of participants with treatment-emergent adverse events grouped in categories regarding relationship to study drug as assessed by the investigator, serious or life-threatening as assessed by the investigator, participants who died or their event led to withdrawal from study, and participants who experienced thrombotic or thromboembolic AEs.
Time Frame: Day 1 to up to Month 9
Population: Intent to treat population (ITT)
Measure: Number; unit: participants
Arm/Group | Tranexamic Acid
Number analyzed (Participants) | 260
participants
  Any treatment-emergent AE | 218
  Definitely related AE | 1
  Probably related AE | 3
  Possibly related AE | 60
  Serious AE | 5
  Life-threatening AE | 2
  Died | 0
  AE led to withdrawal from study | 6
  Thrombotic or thromboembolic AE | 0

2. Secondary Outcome: Participants With Abnormal Gynecological Examinations
Description: Participants with abnormal gynecological examination findings based on endometrial biopsies and transvaginal ultraonogrphy (TVU) are summarized. Clinically significant results from the endometrial biopsies are results that are not benign. Abnormalities found during transvaginal ultrasonography (TVU) are detailed in the AE listings. Please refer to AE listings.
Time Frame: Day 1 to up to Month 9
Population: Intent to treat population
Measure: Number; unit: participants
Arm/Group | Tranexamic Acid
Number analyzed (Participants) | 260
participants
  Significant results from endometrial biopsies | 0
  Abnormalities noted on TVU | 3
  Discontinued due to failed physical exam | 0

3. Secondary Outcome: Mean Blood Pressure Measurements at Week 36
Description: Mean systolic and diastolic blood pressure measurements taken at week 36
Time Frame: approximately week 36
Population: Intent to treat population of participants with week 36 blood pressure data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Tranexamic Acid
Number analyzed (Participants) | 200
mmHg
  Systolic blood pressure | 118.94 (14.272)
  Diastolic blood pressure | 75.09 (10.167)

4. Secondary Outcome: Participants With Treatment Emergent Adverse Experiences (TEAE) of Laboratory Values Related to Treatment
Description: Participants whose laboratory examinations (hematology, blood chemistry and urinalysis) were considered by the investigator to be treatment emergent adverse experiences (TEAE) and related to treatment. Also indicated is whether the TEAE lab parameter caused the participant to discontinue from the study.
Time Frame: Day 1 to up to Month 9
Population: Intent to treat population
Measure: Number; unit: participants
Arm/Group | Tranexamic Acid
Number analyzed (Participants) | 260
participants
  Hematology TEAE related to study drug | 1
  Discontinued due to hematology TEAE | 1
  Blood chemistry TEAE related to study drug | 1
  Discontinued due to blood chemistry TEAE | 0
  Urinalysis TEAE related to study drug | 2
  Discontinued due to urinalysis TEAE | 0

5. Secondary Outcome: Mean Intraocular Pressure at Month 9
Description: Mean intraocular pressure at month 9 or the early termination visit.
Time Frame: Day 1 up to Month 9
Population: Intent to treat participants who had ophthalmic exams.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Tranexamic Acid
Number analyzed (Participants) | 199
mmHg
  Right eye | 15.4 (2.866)
  Left eye | 15.3 (2.797)

6. Secondary Outcome: Mean Fridericia-corrected QT Interval (QTcFRI) at Month 9
Description: The QT interval is the period that extends from the beginning of ventricular depolarization until the end of ventricular repolarization
Time Frame: Month 9
Population: Intent to treat participants who had an electrocardiogram (ECG) at month 9
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Tranexamic Acid
Number analyzed (Participants) | 193
milliseconds | 412.3 (15.896)

ADVERSE EVENTS:
Time Frame: Treatment-emergent AEs: day 1 up to month 9
Arm/Group | Tranexamic Acid
Serious Adverse Events (participants affected / at risk) | 5/260
Other Adverse Events (participants affected / at risk) | 218/260
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tranexamic Acid (N=260)
Blood glucose decreased (Investigations) | 1
Carcinoid tumour of the stomach (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Brain stem infarction (Nervous system disorders) | 1
Intracranial aneurysm (Nervous system disorders) | 1
Trigeminal neuralgia (Nervous system disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tranexamic Acid (N=260)
Anaemia (Blood and lymphatic system disorders) | 10
Ear congestion (Ear and labyrinth disorders) | 1
Ear discomfort (Ear and labyrinth disorders) | 1
Ear pain (Ear and labyrinth disorders) | 4
Ear pruritus (Ear and labyrinth disorders) | 1
Tympanic membrane disorder (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 3
Hypothyroidism (Endocrine disorders) | 1
Chalazion (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 1
Corneal pigmentation (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Eye discharge (Eye disorders) | 1
Eye irritation (Eye disorders) | 1
Ocular hypertension (Eye disorders) | 1
Retinal artery stenosis (Eye disorders) | 1
Retinal pigmentation (Eye disorders) | 1
Vision blurred (Eye disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 15
Abdominal pain (Gastrointestinal disorders) | 12
Abdominal pain lower (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 15
Anal polyp (Gastrointestinal disorders) | 3
Chapped lips (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 9
Diarrhoea (Gastrointestinal disorders) | 19
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 9
Flatulence (Gastrointestinal disorders) | 2
Food poisoning (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4
Gingival pain (Gastrointestinal disorders) | 1
Gingival swelling (Gastrointestinal disorders) | 1
Lip blister (Gastrointestinal disorders) | 1
Loose stools (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 17
Oesophagitis (Gastrointestinal disorders) | 1
Tongue disorder (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 11
Vomiting (Gastrointestinal disorders) | 6
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 1
Chills (General disorders) | 4
Cyst (General disorders) | 1
Fatigue (General disorders) | 14
Influenza like illness (General disorders) | 15
Localized oedema (General disorders) | 1
Oedema (General disorders) | 2
Pyrexia (General disorders) | 4
Swelling (General disorders) | 2
Cholecystitis (Hepatobiliary disorders) | 1
Multiple allergies (Immune system disorders) | 13
Seasonal allergies (Immune system disorders) | 9
Acute sinusitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 5
Cystitis (Infections and infestations) | 3
Ear infection (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Influenza (Infections and infestations) | 4
Kidney infection (Infections and infestations) | 1
Laryngitis (Infections and infestations) | 2
Onychomycosis (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Pharyngitis streptococcal (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 1
Recurring skin boils (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 4
Salpingitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 22
Tonsillitis (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 9
Urinary tract infection (Infections and infestations) | 8
Vaginal candidiasis (Infections and infestations) | 5
Viral upper respiratory tract infection (Infections and infestations) | 31
Vulvovaginitis trichomonal (Infections and infestations) | 2
Arthropod sting (Injury, poisoning and procedural complications) | 1
Back injury (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Joint injury (Injury, poisoning and procedural complications) | 4
Joint sprain (Injury, poisoning and procedural complications) | 1
Muscle strain (Injury, poisoning and procedural complications) | 2
Post procedural complication (Injury, poisoning and procedural complications) | 1
Post procedural discomfort (Injury, poisoning and procedural complications) | 2
Post procedural pain (Injury, poisoning and procedural complications) | 7
Aspartate aminotransferase increased (Investigations) | 1
Biopsy breast (Investigations) | 1
Blood cholesterol increased (Investigations) | 1
Blood glucose increased (Investigations) | 1
Blood triglycerides increased (Investigations) | 1
Blood urine present (Investigations) | 2
Cardiac murmur (Investigations) | 1
Electrocardiogram T wave abnormal (Investigations) | 1
Faecal occult blood (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 2
Haematocrit decreased (Investigations) | 3
Haemoglobin decreased (Investigations) | 4
Human papilloma virus serology test negative (Investigations) | 1
Human papilloma virus serology test positive (Investigations) | 1
Lipids increased (Investigations) | 2
Lymph node palpable (Investigations) | 1
Mean cell haemoglobin decreased (Investigations) | 1
Monocyte count decreased (Investigations) | 1
Red blood cell count decreased (Investigations) | 1
Serum ferritin decreased (Investigations) | 2
Smear cervix abnormal (Investigations) | 7
Thyroxine increased (Investigations) | 1
Ultrasound uterus (Investigations) | 2
Urinary occult blood positive (Investigations) | 2
Weight increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Insulin resistance (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 15
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 60
Buttock pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1
Muscle cramp (Musculoskeletal and connective tissue disorders) | 11
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 15
Myalgia (Musculoskeletal and connective tissue disorders) | 7
Neck pain (Musculoskeletal and connective tissue disorders) | 13
Pain in extremity (Musculoskeletal and connective tissue disorders) | 20
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 2
Tendonitis (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 114
Migraine (Nervous system disorders) | 20
Paraesthesia (Nervous system disorders) | 3
Restless leg syndrome (Nervous system disorders) | 2
Sedation (Nervous system disorders) | 2
Sinus headache (Nervous system disorders) | 17
Tension headache (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 7
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 1
Depressed mood (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 9
Insomnia (Psychiatric disorders) | 11
Irritability (Psychiatric disorders) | 4
Mood swings (Psychiatric disorders) | 4
Stress symptoms (Psychiatric disorders) | 3
Bladder pain (Renal and urinary disorders) | 1
Cystitis interstitial (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Polyuria (Renal and urinary disorders) | 1
Adenomyosis (Reproductive system and breast disorders) | 1
Breast cyst (Reproductive system and breast disorders) | 2
Breast discharge (Reproductive system and breast disorders) | 1
Breast discomfort (Reproductive system and breast disorders) | 1
Breast mass (Reproductive system and breast disorders) | 1
Breast pain (Reproductive system and breast disorders) | 1
Breast tenderness (Reproductive system and breast disorders) | 5
Cervical polyp (Reproductive system and breast disorders) | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 5
Fibrocystic breast disease (Reproductive system and breast disorders) | 1
Menometrorrhagia (Reproductive system and breast disorders) | 1
Menstrual discomfort (Reproductive system and breast disorders) | 3
Menstrual disorder (Reproductive system and breast disorders) | 1
Nipple pain (Reproductive system and breast disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1
Ovulation pain (Reproductive system and breast disorders) | 1
Paraesthesia of genital female (Reproductive system and breast disorders) | 8
Pelvic pain (Reproductive system and breast disorders) | 2
Premenstrual syndrome (Reproductive system and breast disorders) | 2
Pruritus genital (Reproductive system and breast disorders) | 6
Uterine enlargement (Reproductive system and breast disorders) | 1
Uterine leiomyoma (Reproductive system and breast disorders) | 1
Uterine pain (Reproductive system and breast disorders) | 1
Vaginal discharge (Reproductive system and breast disorders) | 7
Vaginal odour (Reproductive system and breast disorders) | 1
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 4
Asthma exercise induced (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 12
Dry throat (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 9
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 16
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 3
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 6
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 2
Acne (Skin and subcutaneous tissue disorders) | 3
Cold sweat (Skin and subcutaneous tissue disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Lichenification (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 3
Urticaria (Skin and subcutaneous tissue disorders) | 1
Benign breast lump removal (Surgical and medical procedures) | 1
Meniscus operation (Surgical and medical procedures) | 1
Surgery (Surgical and medical procedures) | 1
Flushing (Vascular disorders) | 1
Hypertension (Vascular disorders) | 3
Hypotension (Vascular disorders) | 1
Varicose vein (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.